CLINICAL TRIAL: NCT01295125
Title: Randomized Control Trial of Biologic Mesh (XenMATRIXTM) vs. Component Separation Alone in Contaminated Ventral Hernia Repair:a Pilot Study
Brief Title: Comparative Study of Biologic Mesh Versus Repair With Component Separation.
Acronym: Davol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor chose not to move forward with study
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Bard Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-10-23
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Ventral Hernia
Keywords: Infected ventral hernia; Contaminated incisional hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- XenMATRIX (Experimental): Use of XenMATRIX mesh to repair hernia
  Interventions: Device: XenMATRIX mesh; Procedure: Open abdominal ventral hernia repair

INTERVENTIONS:
Device: XenMATRIX mesh — Use of XenMATRIX mesh in the repair of contaminated ventral hernia repair
  Other Names: Davol Biologic mesh
Procedure: Open abdominal ventral hernia repair — Abdominal ventral hernia repair with native tissue
  Other Names: Abdominal ventral hernia repair with native tissue

SUMMARY:
The purpose of this study is to compare open abdominal incisional hernia repair using XenMATRIX biologic mesh versus repair with their own tissue. This study will provide information in determining if a biological mesh is necessary to provide a sturdy repair for a ventral hernia.

DETAILED DESCRIPTION:
This study will involve comparison of open abdominal incisional hernia repair with XenMATRIX biologic graft versus repair with native tissue.

The current study seeks to evaluate XenMATRIXTM, an FDA approved biologic graft for repairing contaminated abdominal wall defects.

This study will provide significant insight for the reconstructive surgeon and patient to determine whether a biologic graft is necessary for the reconstruction of a contaminated ventral hernia repair to provide a durable single staged repair.

ELIGIBILITY:
Inclusion Criteria:

1. Is an adult ≥ 18 years old of either gender
2. Will undergo a planned open abdominal incisional hernia repair
3. Has a defect that can be repaired primarily without tension with myofascial advancement flaps and requires no more than 1 piece of surgical mesh (largest mesh size (19 x 35 cm)
4. Contamination is known preoperatively, e.g. repair in the presence of a chronic wound, the presence of a stoma or in conjunction with a bowel resection, or such contaminations occurs intraoperatively, e.g. inadvertent enterotomy or opening of other hollow intra-abdominal viscus
5. Infection is known due to local frank signs of incisional drainage, fistula formation or abdominal abscess following prior surgical abdominal surgery or presence of infected mesh
6. Has an estimated hernia size of ≥ 3cm to 20cm in maximal width by physical exam
7. Is considered a clean-contaminated or contaminated case per Surgical Site Infection Risk Guidelines
8. Is willing and able to return for all scheduled and required study visits
9. Is willing and able to provide written informed consent for study participation

Exclusion Criteria:

1. Has a defect that the surgeon cannot achieve primary fascial apposition and requires a bridge of mesh
2. Is a clean or dirty case per Surgical Site Infection Risk Guidelines
3. Has conditions that would adversely affect subject safety as per product labeling
4. Will undergo a laparoscopic hernia repair
5. Has a nidus of chronic colonization, such as chronic indwelling bladder catheter or significant amounts of non-removable infected mesh
6. Has conditions which preclude abdominal imaging at a standard imaging facility
7. Has an anticipated survival of < 24 months
8. Care plan is to perform a staged repair over 45 days
9. Is bedridden or otherwise non-ambulatory (i.e. is unable to independently transfer into and out of a wheelchair)
10. Is ASA class 4 or 5
11. BMI over 45
12. Is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Rosen, MD., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | XenMATRIX
Started | 9
Completed | 0
Not Completed | 9
Not completed — Study stopped prematurely | 9

BASELINE CHARACTERISTICS:
Arm/Group | XenMATRIX
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Postoperative Hernia Recurrence
Time Frame: two years after surgery date
Population: No data collected
Arm/Group | XenMATRIX
Number analyzed (Participants) | 0

2. Secondary Outcome: Compare the Short-term Clinical Outcomes of Postoperative Wound Events
Time Frame: two years after surgery date
Population: No data collected
Arm/Group | XenMATRIX
Number analyzed (Participants) | 0

3. Secondary Outcome: Length of Hospital Stay
Description: Participants will be followed for the duration of the hospital stay, an expected average of 1 week
Time Frame: Number of days up to 1 week
Population: No data collected
Arm/Group | XenMATRIX
Number analyzed (Participants) | 0

4. Secondary Outcome: Length of Resource Utilization
Time Frame: two years after surgery date
Population: No data collected
Arm/Group | XenMATRIX
Number analyzed (Participants) | 0

5. Secondary Outcome: Antibiotic Usage and Days
Time Frame: two years after surgery date
Population: No data collected
Arm/Group | XenMATRIX
Number analyzed (Participants) | 0

6. Secondary Outcome: Resumption of Activities of Daily Living
Time Frame: two years after surgery date
Population: No data collected
Arm/Group | XenMATRIX
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AE data not collected
Description: AE data not collected
Arm/Group | XenMATRIX
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No